CLINICAL TRIAL: NCT02458729
Title: The Blood Saving Effect and Wound-related Complications of Tranexamic Acid in Mininally Invasive Total Knee Arthroplasty With Rivaroxaban as Thromboprophylaxis
Brief Title: The Blood Saving Effect of Tranexamic Acid in Total Knee Arthroplasty With Rivaroxaban as Thromboprophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Jun-Wen, Clinical Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NMRPG8B6181
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Tranexamic Acid; Total Knee Arthroplasty; Rivaroxaban
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tranexamic Acid; Tranylcypromine; Saline Solution; Sodium Chloride; Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Group (Placebo Comparator): Primary total knee replacement with 0.9% normal saline 20ml administration intravenously twice, five minutes before deflation of the tourniquet and 3 hours after operation Oral rivaroxaban (10mg) QD on PostOp Day 1 to 14 for VTE prophylaxis
  Interventions: Drug: 0.9% Normal Saline (intraoperative); Drug: 0.9% Normal Saline (3 hours after operation); Drug: rivaroxaban (10mg)
- One-dose TXA Group (Active Comparator): Primary total knee replacement with 1 g Tranexamic Acid 5%,5ml/amp administrated intravenously five minutes before deflation of the tourniquet. and then 0.9% normal saline 20ml administration intravenously 3 hours after operation Oral rivaroxaban (10mg) QD on PostOp Day 1 to 14 for VTE prophylaxis
  Interventions: Drug: Tranexamic Acid 5%,5ml/amp (intraoperative); Drug: 0.9% Normal Saline (3 hours after operation); Drug: rivaroxaban (10mg)
- Two-dose TXA Group (Active Comparator): Primary total knee replacement with 1 g Tranexamic Acid 5%,5ml/amp administrated intravenously twice, five minutes before deflation of the tourniquet and 3 hours after operation Oral rivaroxaban (10mg) QD on PostOp Day 1 to 14 for VTE prophylaxis
  Interventions: Drug: Tranexamic Acid 5%,5ml/amp (intraoperative); Drug: Tranexamic Acid 5%,5ml/amp (3 hours after operation); Drug: rivaroxaban (10mg)

INTERVENTIONS:
Drug: Tranexamic Acid 5%,5ml/amp (intraoperative) — tranexamic acid 1g administered intravenously five minutes before deflation of the tourniquet
  Other Names: Transamine
  Arms: One-dose TXA Group; Two-dose TXA Group
Drug: Tranexamic Acid 5%,5ml/amp (3 hours after operation) — tranexamic acid 1g administered intravenously 3 hours after operation
  Other Names: Transamine
  Arms: Two-dose TXA Group
Drug: 0.9% Normal Saline (intraoperative) — 0.9% Normal Saline 20ml administered intravenously five minutes before deflation of the tourniquet
  Other Names: 0.9% sodium chloride
  Arms: Placebo Group
Drug: 0.9% Normal Saline (3 hours after operation) — 0.9% Normal Saline 20ml administered intravenously 3 hours after operation
  Other Names: 0.9% Normal Saline
  Arms: One-dose TXA Group; Placebo Group
Drug: rivaroxaban (10mg) — Oral rivaroxabam (10mg) QD on PostOp Day 1 to 14
  Other Names: Xarelto

SUMMARY:
The aim of this study was to conduct a prospective, randomized, double-blind study and assess the efficacy of and safety for thromboprophylaxis of rivaroxaban in total knee arthroplasty patients when tranexamic acid is used for bleeding prophylaxis.

DETAILED DESCRIPTION:
Total knee arthroplasty is an effective procedure for end-stage arthritis of the knee in terms of pain relief and functional recovery. However, this procedure is associated with a substantial perioperative blood loss. As high as 69% allogeneic blood transfusion rate was reported in patients receiving total knee arthroplasty when preoperative haemoglabin level was <13 g/dl. Tranexamic acid (TXA), an antifibrinolytic, given intraoperatively, has been reported to be effective in reducing one third of postoperative blood loss in standard total knee arthroplasty. Our previous study showed that TXA reduced total blood loss from 1453mL to 833mL (p<0.001) and the need for transfusion from 20% to 4% (p=0.014) in total knee patients with enoxaparin (Clexane; Glaxo-Smith-Kline, Brentford, United Kindom) for thromboprophylaxis.

In recent years, there have been more effective and practical methods for thrombophylaxis in total hip and knee replacement surgeries. Rivaroxaban is one of the first oral factor Xa inhibitors licensed for this regard. The advantages of rivaroxaban include oral administration, no need to monitor blood levels and no dosing adjustments which are convenient for short hospital stay in contemporary total knee arthroplasty. Its efficacy in preventing venous thromboembolism (VTE) after total knee arthroplasty have been extensitvely investigated in RECORD (Regulation of Coagulation in Orthopaedic surgery to prevent Deep-vein thrombosis and pulmonary embolism) 3 and 4 studies, and the results showed that rivaroxaban 10mg once daily was superior to enoxaparin 40mg subcutaneously once daily or 30mg every 12 hours for 10 to 14 days. Despite of its clinical efficacy in VTE prophylaxis, orthopaedic surgeons are still sceptic in routine use of rivaroxaban in knee and hip surgery and concerned about the increased risk of bleeding complications. A higher reoperation rate regarding wound complications within 30 days of hip and knee replacement in the rivaroxaban group than the tinzaparin group (2.94% versus 1.8%) was reported recently. Similar event has been reported in other studies. However, all these studies did not use TXA as bleeding prophylaxis after hip and knee replacement surgery. The risk of increasing VTE by use of TXA, owing to its antifibrinolytic effects, is the cause of concern.

The aim of this study was to conduct a prospective, randomized, double-blind study and assess the efficacy of and safety for thromboprophylaxis of rivaroxaban in total knee arthroplasty patients when TXA is used for bleeding prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* End-stage arthritis of the knee
* Failure of medical treatment or rehabilitation
* Hemoglobin > 10g/dl
* No use of non-steroid anti-inflammatory agent one week before operation

Exclusion Criteria:

* Preoperative Hemoglobin ≦10 g/dl
* History of infection or intraarticular fracture of the affective knee
* Renal function deficiency (GFR < 55 ml/min/1.73m2)which is relative contraindicated for venography
* Elevated liver enzyme, history of liver cirrhosis, impaired liver function and coagulopathy (including long-term use anticoagulant)
* History of deep vein thrombosis, ischemic heart disease or stroke

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence of any deep-vein thrombosis, non-fatal pulmonary embolism, or all-cause mortality | within 15 days after surgery (2 days after the last dose of rivaroxaban )
  Primary efficacy outcome is the composite of any deep-vein thrombosis, non-fatal pulmonary embolism, or all-cause mortality
Incidence of major bleeding after the first dose of rivaroxaban and all death related to postoperative bleedings | within 15 days after surgery (2 days after the last dose of rivaroxaban )
  Primary safety outcome is the composite of major bleeding after the first dose of rivaroxaban and all death related to postoperative bleedings. Major bleeding was defined as bleeding that was fatal, that involved a critical organ, or that required reoperation or clinically overt bleeding outside the surgical site that was associated with a decrease in the hemoglobin level of 2 g or more per deciliter or requiring infusion of 2 or more units of blood

SECONDARY OUTCOMES:
Incidence of major venous thromboembolism | within 15 days after surgery (2 days after the last dose of rivaroxaban
  The secondary efficacy outcomes include major venous thromboemolism defined as the composite of proximal deep-vein thrombosis, non-fatal pulmonary embolism, and VTE related death
Secondary safety outcome was composite of any non-major bleeding and all wound complications after operation | within 15 days after surgery (2 days after the last dose of rivaroxaban
  Non-major bleeding including hemorrhagic wound complications (excessive wound hematoma or bleeding at the surgical site
Incidence of wound complications after surgery | within 30 days of the procedure
  composite of hematoma, superficial wound infection, and deep infection requiring return to surgery
Total blood loss after surgery | From the operation to the postoperative day 4
  Total blood loss was calculated according to Nadler et al., which used maximum postoperative reduction of the Hb level adjust for weight and height of the patient. The formula is as follows, Total blood loss = (Total blood volume x [change in Hb level / preoperative Hb level])x1000+volume transfused

OTHER OUTCOMES:
Incidence of venographic positive deep-vein thrombosis (any, proximal, distal) | on the second day after last dose of rivaroxaban (POD 15)
Incidence of positive finding of pulmonary embolism by computed tomography | on the second day after last dose of rivaroxaban (POD 15)
  In case of suspected pulmonary embolism, computed tomography of the chest was performed

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Wen Wang, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Koahsiung, Taiwan, Taiwan

REFERENCES:
- [Background] Petaja J, Myllynen P, Myllyla G, Vahtera E. Fibrinolysis after application of a pneumatic tourniquet. Acta Chir Scand. 1987 Nov-Dec;153(11-12):647-51. PMID 3124428
- [Background] Kambayashi J, Sakon M, Yokota M, Shiba E, Kawasaki T, Mori T. Activation of coagulation and fibrinolysis during surgery, analyzed by molecular markers. Thromb Res. 1990 Oct 15;60(2):157-67. doi: 10.1016/0049-3848(90)90294-m. PMID 2149215
- [Background] Hiippala S, Strid L, Wennerstrand M, Arvela V, Mantyla S, Ylinen J, Niemela H. Tranexamic acid (Cyklokapron) reduces perioperative blood loss associated with total knee arthroplasty. Br J Anaesth. 1995 May;74(5):534-7. doi: 10.1093/bja/74.5.534. PMID 7772427
- [Background] Bierbaum BE, Callaghan JJ, Galante JO, Rubash HE, Tooms RE, Welch RB. An analysis of blood management in patients having a total hip or knee arthroplasty. J Bone Joint Surg Am. 1999 Jan;81(1):2-10. doi: 10.2106/00004623-199901000-00002. PMID 9973048
- [Background] Tanaka N, Sakahashi H, Sato E, Hirose K, Ishima T, Ishii S. Timing of the administration of tranexamic acid for maximum reduction in blood loss in arthroplasty of the knee. J Bone Joint Surg Br. 2001 Jul;83(5):702-5. doi: 10.1302/0301-620x.83b5.11745. PMID 11476309
- [Background] Prevention of venous thromboembolism. International Consensus Statement (guidelines according to scientific evidence). Int Angiol. 1997 Mar;16(1):3-38. No abstract available. PMID 9165356
- [Background] Clagett GP, Anderson FA Jr, Geerts W, Heit JA, Knudson M, Lieberman JR, Merli GJ, Wheeler HB. Prevention of venous thromboembolism. Chest. 1998 Nov;114(5 Suppl):531S-560S. doi: 10.1378/chest.114.5_supplement.531s. No abstract available. PMID 9822062
- [Background] Turpie AG, Lassen MR, Davidson BL, Bauer KA, Gent M, Kwong LM, Cushner FD, Lotke PA, Berkowitz SD, Bandel TJ, Benson A, Misselwitz F, Fisher WD; RECORD4 Investigators. Rivaroxaban versus enoxaparin for thromboprophylaxis after total knee arthroplasty (RECORD4): a randomised trial. Lancet. 2009 May 16;373(9676):1673-80. doi: 10.1016/S0140-6736(09)60734-0. Epub 2009 May 4. PMID 19411100
- [Background] Lassen MR, Ageno W, Borris LC, Lieberman JR, Rosencher N, Bandel TJ, Misselwitz F, Turpie AG; RECORD3 Investigators. Rivaroxaban versus enoxaparin for thromboprophylaxis after total knee arthroplasty. N Engl J Med. 2008 Jun 26;358(26):2776-86. doi: 10.1056/NEJMoa076016. PMID 18579812
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271
- [Background] Geerts WH, Heit JA, Clagett GP, Pineo GF, Colwell CW, Anderson FA Jr, Wheeler HB. Prevention of venous thromboembolism. Chest. 2001 Jan;119(1 Suppl):132S-175S. doi: 10.1378/chest.119.1_suppl.132s. No abstract available. PMID 11157647
- [Background] Jameson SS, Bottle A, Malviya A, Muller SD, Reed MR. The impact of national guidelines for the prophylaxis of venous thromboembolism on the complications of arthroplasty of the lower limb. J Bone Joint Surg Br. 2010 Jan;92(1):123-9. doi: 10.1302/0301-620X.92B1.22751. PMID 20044690
- [Background] Patel VP, Walsh M, Sehgal B, Preston C, DeWal H, Di Cesare PE. Factors associated with prolonged wound drainage after primary total hip and knee arthroplasty. J Bone Joint Surg Am. 2007 Jan;89(1):33-8. doi: 10.2106/JBJS.F.00163. PMID 17200307
- [Background] Lotke PA. Rivaroxaban for thromboprophylaxis. N Engl J Med. 2008 Nov 13;359(20):2174; author reply 2175-6. No abstract available. PMID 19009675
- [Background] Jensen CD, Steval A, Partington PF, Reed MR, Muller SD. Return to theatre following total hip and knee replacement, before and after the introduction of rivaroxaban: a retrospective cohort study. J Bone Joint Surg Br. 2011 Jan;93(1):91-5. doi: 10.1302/0301-620X.93B1.24987. PMID 21196550
- [Background] Ido K, Neo M, Asada Y, Kondo K, Morita T, Sakamoto T, Hayashi R, Kuriyama S. Reduction of blood loss using tranexamic acid in total knee and hip arthroplasties. Arch Orthop Trauma Surg. 2000;120(9):518-20. doi: 10.1007/s004029900132. PMID 11011672
- [Background] Lin PC, Hsu CH, Chen WS, Wang JW. Does tranexamic acid save blood in minimally invasive total knee arthroplasty? Clin Orthop Relat Res. 2011 Jul;469(7):1995-2002. doi: 10.1007/s11999-011-1789-y. Epub 2011 Feb 1. PMID 21286886
- [Background] Friedman RJ, Gallus AS, Cushner FD, Fitzgerald G, Anderson FA Jr; Global Orthopaedic Registry Investigators. Physician compliance with guidelines for deep-vein thrombosis prevention in total hip and knee arthroplasty. Curr Med Res Opin. 2008 Jan;24(1):87-97. doi: 10.1185/030079908x242746. PMID 18028586
- [Background] Warwick D, Dahl OE, Fisher WD; International Surgical Thrombosis Forum. Orthopaedic thromboprophylaxis: limitations of current guidelines. J Bone Joint Surg Br. 2008 Feb;90(2):127-32. doi: 10.1302/0301-620X.90B2.20106. PMID 18256075
- [Background] Haas SB, Cook S, Beksac B. Minimally invasive total knee replacement through a mini midvastus approach: a comparative study. Clin Orthop Relat Res. 2004 Nov;(428):68-73. doi: 10.1097/01.blo.0000147649.82883.ca. PMID 15534521
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Background] Lin PC, Hsu CH, Huang CC, Chen WS, Wang JW. The blood-saving effect of tranexamic acid in minimally invasive total knee replacement: is an additional pre-operative injection effective? J Bone Joint Surg Br. 2012 Jul;94(7):932-6. doi: 10.1302/0301-620X.94B7.28386. PMID 22733948
- [Background] Jameson SS, Rymaszewska M, Hui AC, James P, Serrano-Pedraza I, Muller SD. Wound complications following rivaroxaban administration: a multicenter comparison with low-molecular-weight heparins for thromboprophylaxis in lower limb arthroplasty. J Bone Joint Surg Am. 2012 Sep 5;94(17):1554-8. doi: 10.2106/JBJS.K.00521. PMID 22832942